CLINICAL TRIAL: NCT06953661
Title: Ultrasound Guided Stellate Ganglion Block in Postural Tachycardia Syndrome: A Randomized Double Blind Sham Placebo-controlled Pilot Study
Brief Title: Ultrasound Guided Stellate Ganglion Block in Postural Tachycardia Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Maria Bombardieri, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 80519
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Postural Tachycardia Syndrome
Keywords: stellate ganglion block; regional anesthesia; nerve block
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Twenty patients will be enrolled, with 10 patients allocated to each study arm (treatment and control).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (stellate ganglion block) (Experimental): Patients will receive an ultrasound guided stellate ganglion block (SGB) with 10 ml of 0.5% ropivacaine.
  Interventions: Procedure: Stellate ganglion block; Drug: Ropivacaine
- Control Group (sham injection with saline) (Sham Comparator): Patients will receive a subcutaneous sham injection with saline. Ultrasound imaging will be used to simulate the guidance process as in the active procedure, maintaining consistency in the procedural experience.
  Interventions: Procedure: Sham injection of saline; Drug: Normal saline

INTERVENTIONS:
Procedure: Stellate ganglion block — Patients will receive a SGB
  Arms: Intervention Group (stellate ganglion block)
Procedure: Sham injection of saline — Patients will receive a subcutaneous sham injection of saline
  Arms: Control Group (sham injection with saline)
Drug: Ropivacaine — The SGB group will receive ropivacaine 0.5% 10ml
  Arms: Intervention Group (stellate ganglion block)
Drug: Normal saline — The control group will receive normal saline in the sham injection.
  Arms: Control Group (sham injection with saline)

SUMMARY:
This single-center study aims to evaluate both immediate and long-term outcomes of stellate ganglion block (SGB) in a cohort of rigorously phenotyped patients with Postural Tachycardia Syndrome (POTS). By assessing the effects of SGB, this study seeks to determine its viability as an intervention for symptom control in POTS.

DETAILED DESCRIPTION:
Postural Tachycardia Syndrome (POTS) is a heterogeneous condition affecting approximately 0.2% of the global population, predominantly young women of childbearing age. It is characterized by significant functional impairment and a constellation of symptoms, including lightheadedness, cognitive dysfunction, blurred vision, irritability, palpitations, and chest discomfort, which occur upon standing and improve when lying down. Although current pharmacological and non-pharmacological treatments alleviate symptoms for some patients, many remain significantly disabled. These challenges highlight the urgent need for novel treatment strategies, particularly non-pharmacological approaches.

This study is a randomized controlled trial with a control group. The study team will enroll 20 patients with POTS, assigning 10 to the intervention group and 10 to the control group.

The goal of the study is to evaluate the effectiveness of SGB in improving heart rate, markers of sympathetic hyperactivity, and POTS symptoms comparing to a sham saline injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) diagnosed with POTS
* Ability to provide informed consent
* Ability to comply with 3 follow up visits
* English speaking and capable of signing informed consent and complying with protocol requirements

Exclusion Criteria:

* Allergy to local anesthetics
* Severe coagulopathy
* History of or currently being treated for clinically significant ongoing cardiac arrhythmia, heart failure, myocarditis, pulmonary embolism requiring anticoagulation, pulmonary fibrosis or other pulmonary diagnosis that in the investigator's opinion may contribute to symptoms of POTS
* Inability to maintain a stable medication regiment for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-13 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
COMPASS 31 total score | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  The change in Composite Autonomic Symptom Score 31 (COMPASS-31) from baseline to first follow-up visit. The COMPASS-31 scale measures autonomic dysfunctions through 31 patient-reported questions. A higher score indicates worse autonomic dysfunction.

SECONDARY OUTCOMES:
Magnitude of postural tachycardia | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Change in magnitude of postural tachycardia (a heart rate increase within the first 10 minutes of standing) from baseline to first and second follow up visit.
Heart rate variability (HRV) | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Change in heart rate variability (HRV) metrics (time and frequency domains) from baseline to first and second follow up visit
Plasma catecholamine levels | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Measure the change in plasma catecholamine levels from baseline to first and second follow up visits
Survey of Postural Orthostatic Tachycardia Syndrome Symptoms (SPOTS) | Baseline (day -21 to -1 before intervention) to 1-2 weeks, then day 74 to 94 following study intervention
  SPOTS evaluates the frequency and severity of common POTS symptoms, The higher the score, the greater the symptom burden. A reduction in SPOTS score suggests clinical improvement. SPOTS scores at 1st and 2nd FU are compared to baseline SPOTS scores.
VOSS score | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Change in VOSS score at 1st and 2nd FU compared to baseline. The Vanderbilt Orthostatic Symptom Score (VOSS) is a tool used to assess and track the severity of symptoms associated with postural orthostatic tachycardia syndrome (POTS). It helps quantify a patient's symptom burden by having them rate the severity of 9 symptoms (mental clouding, blurred vision, shortness of breath, rapid heartbeat, tremulousness, chest discomfort, headache, lightheadedness, and nausea) on a scale of 0 to 10, where 0 indicates no symptoms.
FSS score | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Change in FSS score at 1st and 2nd FU compared to baseline. The Fatigue Severity Scale (FSS) is a questionnaire used to measure the severity of fatigue and its impact on daily activities. It's a 9-item scale where respondents rate their agreement with statements about fatigue using a 7-point scale, with 1 being "strongly disagree" and 7 being "strongly agree". The total FSS score is calculated by summing the responses, with a higher score indicating greater fatigue severity.
PROMIS Cognitive Function Short Form 6a | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Change in the PROMIS Cognitive Function Short Form 6a score at 1st and 2nd FU compared to baseline. Short Form 6a is a six-item sub-set scale of the PROMIS (Patient Reported Outcomes Measurement Information System) Cognitive Function item bank that assesses patient-perceived cognitive deficits. The questions use a 5-point response scale, ranging from "Not at all" to "Very much". A higher score generally indicates better perceived cognitive ability.
EQ-5D score | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Change in EQ-5D score at 1st and 2nd FU compared to baseline. The EQ-5D is a questionnaire for measuring patient-reported outcomes which assesses health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D index score ranges from 0 to 1, where 1 represents perfect health, 0 represents a state as bad as death, and values between 0 and 1 represent different levels of health, with higher values indicating better health.
PGI-S rating | Baseline (day -21 to -1 before intervention)
  The PGI-S (Patient Global Impression of Severity) is a single-item, 7-point scale used to assess a patient's perception of the current severity of their condition. A rating of 1 indicates "normal, not at all ill," while a rating of 7 indicates "among the most extremely ill patients." This self-reported measure provides a global assessment of illness severity from the patient's perspective and is commonly used in clinical trials to gauge baseline condition or monitor progression over time.
PGI-C rating | First follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  The PGI-C (Patient Global Impression of Change) is a 7-point scale used to assess a patient's perceived change in their health or condition after an intervention. A rating of 1 indicates "very much improved," while a rating of 7 indicates "very much worse". It's a self-reported measure that reflects a patient's belief about the efficacy of treatment.
CGI-S rating | Baseline (day -21 to -1 before intervention)
  The CGI-S (Clinical Global Impression of Severity) is a 7-point scale used by clinicians to assess the severity of a patient's illness at a given point in time. A rating of 1 indicates "normal, not at all ill," while a rating of 7 indicates "among the most extremely ill patients." This clinician-rated measure provides an overall impression of the patient's current condition, based on clinical judgment and all available information, including patient history, symptoms, and behavior.
CGI-C rating | First follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  The Clinical Global Impression of Change (CGI-C) is a scale used to assess the clinical change or improvement in a patient's condition over time. CGI-C scores range from 1 (very much improved) through to 7 (very much worse).
BAI score | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Reduction in anxiety and depression symptoms as measured by the BAI score. Beck Anxiety Inventory (BAI) is a 21-item self-report questionnaire designed to assess the severity of anxiety symptoms. Each item is rated on a 4-point scale (0 = not at all to 3 = severely). The total score ranges from 0 to 63. Higher scores indicate greater severity of anxiety symptoms.
BDI score | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Reduction in anxiety and depression symptoms as measured by the BDI score. Beck Depression Inventory (BDI) is a 21-question multiple-choice self-report inventory for measuring the severity of depression. The total score ranges from 0 to 63. Higher total scores indicate more severe depressive symptoms.
Adrenergic G-protein-coupled receptor autoantibody activity | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Measure the change in adrenergic G-protein-coupled receptor autoantibody concentrations from baseline to first and second follow up visits from stored serum samples.
Inflammatory markers (including but not limited to IL1, IL6, IL8, TNF) | Baseline (day -21 to -1 before intervention), first follow-up (day 1 to 21 after the intervention) and second follow-up (day 74 to 94 after the intervention)
  Measure the change in inflammatory markers concentrations (including but not limited to IL1, IL6, IL8, TNF) from baseline to first and second follow up visits from stored serum samples
Horner's syndrome | Within 10 minutes after the procedure
  Proportion of patients achieving Horner's syndrome post-SGB as a measure of block success
Facial skin temperature | Within 10 minutes after the procedure
  Measure the change in facial skin temperature (C°) post-procedure
Facial sweating | Within 10 minutes after the procedure
  Sweat testing will be performed following the procedure. The patient is coated with a moisture-sensitive powder that changes color following the increase in facial blood flow following the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernino S, Bourne KM, Stiles LE, Grubb BP, Fedorowski A, Stewart JM, Arnold AC, Pace LA, Axelsson J, Boris JR, Moak JP, Goodman BP, Chemali KR, Chung TH, Goldstein DS, Diedrich A, Miglis MG, Cortez MM, Miller AJ, Freeman R, Biaggioni I, Rowe PC, Sheldon RS, Shibao CA, Systrom DM, Cook GA, Doherty TA, Abdallah HI, Darbari A, Raj SR. Postural orthostatic tachycardia syndrome (POTS): State of the science and clinical care from a 2019 National Institutes of Health Expert Consensus Meeting - Part 1. Auton Neurosci. 2021 Nov;235:102828. doi: 10.1016/j.autneu.2021.102828. Epub 2021 Jun 5. PMID 34144933
- [Background] Doherty TA, White AA. Postural orthostatic tachycardia syndrome and the potential role of mast cell activation. Auton Neurosci. 2018 Dec;215:83-88. doi: 10.1016/j.autneu.2018.05.001. Epub 2018 May 4. PMID 30033040
- [Background] Duricka D, Liu L. Reduction of long COVID symptoms after stellate ganglion block: A retrospective chart review study. Auton Neurosci. 2024 Aug;254:103195. doi: 10.1016/j.autneu.2024.103195. Epub 2024 Jun 13. PMID 38901177
- [Background] Pearson L, Maina A, Compratt T, Harden S, Aaroe A, Copas W, Thompson L. Stellate Ganglion Block Relieves Long COVID-19 Symptoms in 86% of Patients: A Retrospective Cohort Study. Cureus. 2023 Sep 13;15(9):e45161. doi: 10.7759/cureus.45161. eCollection 2023 Sep. PMID 37711269
- [Background] Cha YM, Li X, Yang M, Han J, Wu G, Kapa SC, McLeod CJ, Noseworthy PA, Mulpuru SK, Asirvatham SJ, Brady PA, Rho RH, Friedman PA, Lee HC, Tian Y, Zhou S, Munger TM, Ackerman MJ, Shen WK. Stellate ganglion block and cardiac sympathetic denervation in patients with inappropriate sinus tachycardia. J Cardiovasc Electrophysiol. 2019 Dec;30(12):2920-2928. doi: 10.1111/jce.14233. Epub 2019 Nov 6. PMID 31625219
- [Background] Larsen NW, Stiles LE, Miglis MG. Preparing for the long-haul: Autonomic complications of COVID-19. Auton Neurosci. 2021 Nov;235:102841. doi: 10.1016/j.autneu.2021.102841. Epub 2021 Jul 3. PMID 34265539